CLINICAL TRIAL: NCT03196427
Title: A Phase 2b, Extension Study to Determine the Long-term Safety of Vedolizumab IV in Pediatric Subjects With Ulcerative Colitis or Crohn's Disease
Brief Title: Long-term Safety With Vedolizumab Intravenous (IV) in Pediatric Participants With Ulcerative Colitis (UC) or Crohn's Disease (CD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vedolizumab-2005; 2017-002182-21 (EudraCT Number); U1111-1176-5741 (Other: WHO); 17/NE/0258 (Registry Identifier: NRES); MOH_2017-09-18_000649 (Other: CRS); 2023-507766-35-00 (EU CTIS Number)
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vedolizumab High Dose Group (Experimental): Participants with UC or CD having baseline weight of greater than or equal to (>=) 30 kilogram (kg) will receive vedolizumab 300 mg and participants with UC or CD having baseline weight of less than (<) 30 kg will receive vedolizumab 200 mg, IV infusion, every 8 weeks until vedolizumab IV is commercially available for pediatric indication(s) in the participant's country or until other drug access programs become available (whichever comes first), the participant turns 18 years of age and can be transitioned to commercial drug (up to approximately 8 years).
  Interventions: Drug: Vedolizumab
- Vedolizumab Low Dose Group (Experimental): Participants with UC or CD having baseline weight of >= 30 kg will receive vedolizumab 150 mg and participants with UC or CD having baseline weight of < 30 kg will receive vedolizumab 100 mg IV infusion, every 8 weeks until vedolizumab IV is commercially available for pediatric indication(s) in the participant's country or until other drug access programs become available (whichever comes first), the participant turns 18 years of age and can be transitioned to commercial drug (up to approximately 8 years).
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab intravenous infusion
  Other Names: MLN0002; ENTYVIO; KYNTELES

SUMMARY:
The purpose of this study is to determine the safety profile of long-term vedolizumab IV treatment in pediatric participants with UC or CD.

DETAILED DESCRIPTION:
The drug being tested in this study is called Vedolizumab. Vedolizumab is being tested to treat pediatric participants who have moderately to severely active UC or CD.

This study will look at the long-term safety profile in participants who take vedolizumab IV. Participants will continue receiving the same dose assigned from the parent study MLN0002-2003 [NCT03138655], which will remain blinded until week 40.

The dosing regimen selected for the long-term study is intended to maintain clinical response at the lowest possible exposure.

At the discretion of the investigator, participants receiving the low dose (150 or 100 milligram [mg]) of vedolizumab IV may be escalated to the high dose (300 or 200 mg) if the participants demonstrate disease worsening at 2 consecutive visits (scheduled or unscheduled).

Participants who experience continued disease worsening during the study despite being administered vedolizumab 300 or 200 mg every 8 weeks (Q8W) will be discontinued from the study.

Study duration will be until vedolizumab IV is commercially available for pediatric indication(s) in the participant's country or until other drug access programs become available (whichever comes first), the participant turns 18 years of age and can be transitioned to commercial drug, the participant withdraws from the study, or the sponsor decides to close the study (up to approximately 8 years).

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female with UC or CD and was between 2 to 17 years, inclusive, at the time of randomization for Study MLN0002-2003.

   (Note: A participant remains eligible to participate in this study after they reach 18 years of age if they continue to meet the inclusion criteria and do not meet any exclusion criteria.)
2. Has completed Study MLN0002-2003 and, at Week 22, achieved clinical response as defined by a reduction of partial Mayo score of >=2 points and >=25% from Baseline, or a reduction of the Paediatric Ulcerative Colitis Activity Index (PUCAI) of >=20 points from baseline for participants with UC; or a reduction of the CDAI as defined by a >=70-point decrease from Baseline or a decrease of Pediatric Crohn's Disease Activity Index (PCDAI) of >=15 points for participants with CD.
3. May be receiving a therapeutic dose of the following drugs:

   * Oral 5-aminosalicylic acid (5-ASA) compounds.
   * Oral corticosteroid therapy (prednisone or equivalent steroid at a dose less than or equal to [<=] 50 milligram per day [mg/day]) provided the participant was receiving this medication during prior participation in MLN0002-2003.
   * Topical (rectal) treatment with 5-ASA or corticosteroids.
   * Probiotics (example, Saccharomyces boulardii).
   * Antidiarrheals (example, loperamide, diphenoxylate with atropine) for control of chronic diarrhea.
   * Antibiotics used for the treatment of CD (i.e., ciprofloxacin, metronidazole).
   * Azathioprine (AZA) or 6-mercaptopurine (6-MP) or methotrexate (MTX), provided the participant was receiving this medication during prior participation in MLN0002-2003.
4. The participant's vaccinations are up to date as per inclusion criteria number 10 in MLN0002-2003.

Exclusion Criteria:

1. Is female and is lactating or pregnant.
2. Has hypersensitivity or allergies to vedolizumab or any of its excipients.
3. Has withdrawn from Study MLN0002-2003.
4. Has developed any new unstable or uncontrolled cardiovascular, heart failure moderate to severe (New York Class Association III or IV), pulmonary, hepatic, renal, gastrointestinal (GI), genitourinary, hematological, coagulation, immunological, endocrine/metabolic, neurological, or other medical disorder that, in the opinion of the investigator, would confound the study results or compromise participant safety.
5. Has a positive progressive multifocal leukoencephalopathy (PML) subjective symptom checklist prior to the administration of the first dose of study drug.
6. Currently requires major surgical intervention for UC or CD (example, bowel resection), or is anticipated to require major surgical intervention for UC or CD during the study.
7. Has other serious comorbidities that will limit his or her ability to complete the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Treatment-emergent Adverse Events (TEAEs) | Baseline up to approximately 8 years
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.

SECONDARY OUTCOMES:
Percentage of Participants With UC Meeting Clinical Response Based on Complete Mayo Score at Week 32 | Week 32
  Clinical response is defined as a continued reduction in complete mayo score of >=3 points from baseline (at initiation of MLN0002-2003) and continued decrease in rectal bleeding subscore of >=1 point from baseline, or absolute rectal bleeding subscore of <=1 point. Mayo score is an instrument designed to measure disease activity of UC. It consists of 4 subscores: stool frequency, rectal bleeding, findings on endoscopy and physician rating of disease activity, each graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 12; where higher scores indicate more severe disease.
Percentage of Participants With CD Meeting Clinical Response Based on 50 Percent (%) Reduction in Simple Endoscopic Score for Crohn's Disease (SES-CD) Score at Week 32 | Week 32
  Clinical response is defined as a 50% reduction in SES-CD score on endoscopy compared to the baseline endoscopy (at initiation of MLN0002-2003) and continued reduction in CDAI that is a >=70 point decrease from the baseline Crohn's Disease Activity Index (CDAI) score at the initiation of MLN0002-2003. CDAI is a research tool used to quantify the symptoms of participants with Crohn's disease. SES-CD consists of 3 variables: ulcer size, ulcerated and affected surfaces and presence of narrowing each graded from 0 to 3 with score of 0 means no colonic lesions or mucosal healing, and SES-CD greater than (>) 1 indicates the presence of mucosal lesions.
Time to Major Inflammatory Bowel Disease (IBD) - Related Events | Baseline up to approximately 8 years
  Major IBD-related events included hospitalizations, surgeries, or procedures due to UC and CD.
Change from Baseline in IMPACT-III Total and Subscale Scores at Week 24 and Every 24 weeks, Thereafter up to 8 Years | Baseline up to approximately 8 years
  The IMPACT-III questionnaire is a self-reported measure with 35 closed questions encompassing 6 domains: Bowel Symptoms (7 items), Systemic Symptoms (3 items), Social Functioning (12 items), Body Image (3 items), Treatment/Interventions (3 items), and Emotional Functioning (7 items). The IMPACT-III uses a 5-point Likert scale ranging from 1 to 5 for all answers. The outcome score ranges from 35 to 175, with higher scores suggesting better quality of life.
Height Velocity at Week 48 and Every 48 weeks, Thereafter up to 8 Years | Baseline up to approximately 8 years
  Height velocity (centimeter per year [cm/year]) is the change in height per year.
Change from Baseline in Height at Week 24 and Every 24 Weeks, Thereafter up to 8 Years | Baseline up to approximately 8 years
Change from Baseline in Weight at Week 24 and Every 24 Weeks, Thereafter up to 8 Years | Baseline up to approximately 8 years
Change from Baseline in Body Mass Index (BMI) at Week 24 and Every 24 Weeks, Thereafter up to 8 Years | Baseline up to approximately 8 years
  BMI = Weight (in kilograms)/height^2 (in meters).
Percentage of Participants Achieving Tanner Stage V | Baseline up to approximately 8 years
  Tanner Stage Evaluation is a scale used to evaluate growth parameters standardized for age, sex, and pubertal development. Female pubertal development staged by pubic hair development and breast size; male pubertal development staged by size of the genitalia and development of pubic hair. Rated in 5 stages: stage 1 (no development) to 5 (adult-like development in quantity and size). Tanner stage is assessed at or before age 16 years for females or 17 years for males.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (23):
- United States (9):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of California San Francisco, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Nemours Childrens Specialty Care - Jacksonville, Jacksonville, Florida
  - Children's Center for Digestive Healthcare, Atlanta, Georgia
  - Columbia University Medical Center, New York, New York
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Hopital Necker-Enfants Malades, Paris, Île-de-France Region, France
- Hungary (3):
  - BAZ Megyei Korhaz es Egyetemi Oktatokorhaz, Miskolc, Borsod-Abauj Zemplen county
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged, Csongrád megye
  - Debreceni Egyetem Klinikai Kozpont, Debrecen, Hajdú-Bihar
- Israel (5):
  - The Edmond and Lily Safra Children's Hospital - Sheba Medical Center, Ramat Gan, Tel Aviv
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Schneider Children's Medical Center of Israel, Petach Tiqwa
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Poland (3):
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow, Lesser Poland Voivodeship
  - Gabinet Lekarski Dr. Hab. N. Med. Bartosz Korczowski, Rzeszów, Podkarpackie Voivodeship
  - Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi Osrodek Pediatryczny im Marii Konopnic, Lodz, Łódź Voivodeship
- Kharkiv Regional Clinical Children's Hospital, Kharkiv, Ukraine
- Barts and The London NHS Trust, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/5f6b60394db2bf003ab4a220?idFilter=%5B%22vedolizumab-2005%22%5D